CLINICAL TRIAL: NCT06342687
Title: Has High Compliance With Enhanced Recovery After Surgery (ERAS) Protocol Improved 5-Year Survival? - A Cohort Study of 468 Non-Metastatic Colorectal Cancer Patients
Brief Title: Compliance With ERAS and Five Year Survival After Colorectal Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Mateusz Rubinkiewicz, MD PhD, Jagiellonian University
Other Study IDs: JagiellonianU 1
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; ERAS
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: with a compliance rate with ERAS below 80%
- Group 2: with a compliance rate with ERAS of 80% or above
  Interventions: Procedure: High compliance with ERAS protocol

INTERVENTIONS:
Procedure: High compliance with ERAS protocol — Patients were categorized into two groups based on their adherence to the ERAS protocol: group 1 with a compliance rate below 80% and group 2 with a compliance rate of 80% or above.
  Groups: Group 2

SUMMARY:
The Enhanced Recovery after Surgery (ERAS) protocol has transformed perioperative care, representing a significant paradigm shift in managing colorectal cancer patients. While the immediate benefits of Enhanced Recovery After Surgery (ERAS) in expediting postoperative recovery are well-documented and widely acknowledged, it is essential to investigate its long-term implications, particularly its influence on survival rates. The aim of this study will be to analyse the impact of compliance with the ERAS protocol on long- term outcomes after laparoscopic colorectal resection.

DETAILED DESCRIPTION:
The aim of this study will be to analyse the impact of compliance with the ERAS protocol on long- term outcomes after laparoscopic colorectal resection.

The study will be designed as a prospective observational study to compare the long-term effects of surgical treatment of colorectal cancer in two groups of patients: those with high compliance with the ERAS protocol (≥80%) and those with low compliance with the ERAS protocol (<80%).

The primary outcome of the study will be the 5-year survival rate. The inclusion criteria for Group 1 will involve 128 patients with ERAS compliance below 80%. Conversely, Group 2 will consist of 340 patients, all of whom achieved a compliance rate of at least 80%.

The correlation between compliance with the ERAS protocol and 5-year survival will be assessed using the Kaplan-Meier method with log-rank tests. Additionally, survival analysis will be conducted separately for groups with varying cancer stages.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing treatment for colorectal cancer

Exclusion Criteria:

* primary open or emergency surgery,
* transanal endoscopic microsurgery (TEM),
* stage IV of the disease according to the American Joint Committee on Cancer (AJCC) classification,
* multivisceral resection,
* concomitant inflammatory bowel diseases,
* intensive care unit stay immediately after surgery
* lost-to-follow-up patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be divided into two groups based on ERAS protocol compliance. Group 1 comprised patients with adherence below 80%, while Group 2 consisted of individuals who maintained adherence levels of no less than 80%. We established this threshold based on the compliance target set in our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Post operative 5 year survival rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No